CLINICAL TRIAL: NCT00953693
Title: Patient Specific Induced Pluripotency Stem Cells (PSiPS)
Status: Completed | Type: Observational
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: Royan-iPS-001
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2010-04

CONDITIONS: Hepatic Disorders; Eye Disorders
Keywords: Induced pluripotent stem cells; Hepatic disorders; Eye disorders; Blood groups
MeSH Terms: conditions — Digestive System Diseases; Eye Diseases | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Biopsy — Skin biopsy

SUMMARY:
Induced pluripotent stem cells (iPSCs) are adult cells that have been genetically reprogrammed to an embryonic stem cell-like state by being forced to express genes and factors important for maintaining the defining properties of embryonic stem cells. The reprogramming of adult cells into embryonic stem (ES) cells enables the generation of patient-specific stem cells and thus has enormous potential for the treatment and analysis of degenerative diseases. In this project the investigators are going to induce pluripotent stem cells from cell cultures from skin biopsies of patients. The iPS cells will be developed for modeling diseases and drug discovery as well as basic research.

DETAILED DESCRIPTION:
iPS cells are typically derived by transfection of certain stem cell-associated genes into non-pluripotent cells, such as adult fibroblasts. Transfection is typically achieved through viral vectors, such as retroviruses. Transfected genes include the master transcriptional regulators Oct-3/4 (Pouf51) and Sox2, although to enhance the efficiency of induction some other genes e.g. Klf4, c-Myc. In this study after separation the fibroblasts from patient's skin biopsy, the cells are transfected with 4 Yamanaka factors (human Oct4, Sox2, Klf4, c-Myc) after 3-4 weeks, transfected cells are isolated through morphological selection.

ELIGIBILITY:
Inclusion Criteria:

* Donors suffering from different (specified) metabolic disorders
* Donors suffering from different (specified) eye disorders which resulted to blindness
* Special blood group: O Bombay

Exclusion Criteria:

* None

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient who suffering from metabolic disorders
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Royan Institute; Hossein Baharvand, PhD, Study Director — Royan Institute
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- [Result] Seifinejad A, Taei A, Totonchi M, Vazirinasab H, Hassani SN, Aghdami N, Shahbazi E, Yazdi RS, Salekdeh GH, Baharvand H. Generation of human induced pluripotent stem cells from a Bombay individual: moving towards "universal-donor" red blood cells. Biochem Biophys Res Commun. 2010 Jan 1;391(1):329-34. doi: 10.1016/j.bbrc.2009.11.058. Epub 2009 Nov 11. PMID 19912985
- See also: Related Info — http://www.royaninstitute.org